CLINICAL TRIAL: NCT06564415
Title: European Registry for Transperineal Laser Ablation of Prostate (TPLA) for Lower Urinary Tract Symptoms (LUTS) Due to Benign Prostatic Obstruction (BPO)
Brief Title: European Registry for Transperineal Laser Ablation of Prostate (TPLA) for Lower Urinary Tract Symptoms
Status: Recruiting | Type: Observational
Sponsor: University of Florence (Other)
Responsible Party: Principal Investigator, Francesco Sessa, Principal Investigator, University of Florence
Other Study IDs: 25691
Record Dates: First submitted 2024-08-14; First posted 2024-08-21 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Benign Prostatic Hyperplasia; Prostatic Diseases
Keywords: TPLA; Transperineal Laser Ablation; LUTS; BPH; Benign Prostatic Obstruction
MeSH Terms: conditions — Prostatic Hyperplasia; Prostatic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

INTERVENTIONS:
Procedure: Transperineal Laser Ablation of Prostate — Transperineal Laser Ablation of the Prostate is an ultra minimally-invasive procedure that consists in the insertion trough the perineum skin of laser fibers into the prostatic adenoma, under US guidance. Laser energy generates an area of coagulative necrosis that will bring to a reduction of the prostatic volume.

SUMMARY:
The goal of this observational study is to assess mid- and long-term effectiveness of Transperineal Laser Ablation of Prostate (TPLA) for the treatment of lower urinary tract symptoms (LUTS) due to benign prostatic obstruction measured by need and/or time until surgical retreatment.

Data regarding patient-reported outcomes measures (PROMs), flowmetry parameters and safety about consecutive patients undergoing TPLA will be collected in a dedicated platform.

Secondary objectives of the study are:

* To assess functional and safety outcomes in patients treated with transperineal laser ablation for LUTS due to benign prostatic obstruction;
* To identify possible differences in characteristics of patients treated with transperineal laser ablation among the centers and possible relations between treatment application and outcomes, in order to explore the optimal indications and possible limitations of TPLA for LUTS.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years;
* Prostate volume ≥ 30 mL;
* Moderate-to-severe LUTS according to International Prostatic Symptoms Score (IPSS ≥8)
* Consent to participate;

Exclusion Criteria:

* Absence of consent;
* Subsequent withdrawal of consent;
* Diagnosis or suspicion of prostate cancer at multiparametric magnetic resonance
* Documented bladder impaired contractility
* Urethral stenosis
* Previous prostate surgery

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — only biological males can be included
Study Population: Patients referred to the centers participating in the study
Sampling Method: Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2024-01-11 (Actual); Primary Completion 2034-01 (Estimated); Study Completion 2034-01 (Estimated)

PRIMARY OUTCOMES:
Rate of partecipants needing for other surgery | 5 years
  Mid- and long-term effectiveness of TPLA measured by need and/or time until surgical retreatment for BPO (e.g. Transurethral resection of prostate (TURP), endoscopic enucleation, simple prostatectomy)

SECONDARY OUTCOMES:
Number of Participants with Treatment-Related Adverse Events according to Clavien-Dindo Scale | 6 months
  Number of Participants with Treatment-Related Adverse Events as Assessed by Clavien-Dindo scale (score from I to V - higher scores mean a worse outcome)
Number of Participants with Treatment-Related Adverse Events according to Comprehensive Complication Index | 6 months
  Number of Participants with Treatment-Related Adverse Events as Assessed by Comprehensive Complication Index. The Comprehensive Complication Index (CCI) reflects the gravity of the overall complication burden on the patient on a scale from 0 (no complication) to 100 (death)
Change from Baseline in the International Prostatic Symptoms Score (IPSS) | 5 years
  Patient-reported outcome measure about urinary symptoms evaluated by International Prostatic Symptoms Score (IPSS) - values from 0 to 35 (higher scores mean a worse outcome)
Change from Baseline in the IPSS - Quality of Life score | 5 years
  Patient-reported outcome measure about impact of urinary symptoms on quality of life evaluated by IPSS - Quality of Life (QoL) questionnaire (values from 0 to 6 - higher scores mean a worse outcome)
Change from Baseline in the International Index of Erectile Function (IIEF-5) | 5 years
  Patient-reported outcome measure about erectile function evaluated by International Index of Erectile Function (IIEF-5) - values from 0 to 25 (higher values mean a better outcome)
Change from Baseline in the Male Sexual Health Questionnaire bother (MSHQ bother) | 5 years
  Patient-reported outcome measure about impact of ejaculatory disfunctions in quality of life evaluated by Male Sexual Health Questionnaire bother (MSHQ bother) - values from 0 to 5 (higher scores mean a worse outcome)
Change from Baseline in the Male Sexual Health Questionnaire 3-items (MSHQ 3-items) | 5 years
  Patient-reported outcome measure about ejaculatory function evaluated by Male Sexual Health Questionnaire 3-items (MSHQ 3-items) - values from 0 to 15 (higher scores mean a better outcome)
Change from Baseline in maximum flow rate (ml/s) | 5 years
  Change from Baseline in maximum flow rate (ml/s) evaluated at uroflowmetry
Change from Baseline in post void residual volume (ml) | 5 years
  Change from Baseline in post void residual volume (ml) evaluated with sovrapubic ultrasound or bladderscan after spontaneous micturition

CONTACTS AND LOCATIONS:
Locations (1):
- AOU Careggi, Florence, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sessa F, Polverino P, Siena G, Bisegna C, Lo Re M, Spatafora P, Pecoraro A, Rivetti A, Moscardi L, Saladino M, Cocci A, Gacci M, Li Marzi V, Carini M, Minervini A, Campi R, Serni S. Transperineal Laser Ablation of the Prostate (TPLA) for Lower Urinary Tract Symptoms Due to Benign Prostatic Obstruction. J Clin Med. 2023 Jan 19;12(3):793. doi: 10.3390/jcm12030793. PMID 36769454
- [Background] Polverino P, Lo Re M, Saladino M, Pecoraro A, Moscardi L, Rivetti A, Resta GR, Pezzoli M, Romano A, Somani BK, Siena G, Cocci A, Gacci M, Minervini A, Serni S, Campi R, Sessa F. Could transperineal interstitial laser ablation of the prostate be the right option for highly-comorbid patients with lower urinary tract symptoms due to benign prostatic obstruction? A preliminary single-center experience focusing on functional and safety outcomes. Minerva Urol Nephrol. 2024 Oct;76(5):646-649. doi: 10.23736/S2724-6051.23.05479-4. Epub 2023 Dec 13. PMID 38093618
- [Background] Lo Re M, Polverino P, Rivetti A, Pecoraro A, Saladino M, Pezzoli M, Siena G, De Nunzio C, Li Marzi V, Gacci M, Serni S, Campi R, Sessa F. Transperineal laser ablation (TPLA) of the prostate for benign prostatic obstruction: the first 100 patients cohort of a prospective, single-center study. World J Urol. 2024 Jul 10;42(1):402. doi: 10.1007/s00345-024-05077-z. PMID 38985193
- [Background] Canat HL, Gurbuz C, Bozkurt M. Transurethral resection of the prostate (TURP) versus transperineal laser ablation (TPLA) due to benign prostatic hyperplasia (BPH): prospective and comparative study. Int Urol Nephrol. 2023 Nov;55(11):2747-2752. doi: 10.1007/s11255-023-03717-8. Epub 2023 Jul 27. PMID 37498422
- [Background] Minafra P, DE Rienzo G, Gerbasi S, Cindolo L, Battaglia M, Ditonno P. Three years outcomes of transperineal laser ablation of the prostate. Minerva Urol Nephrol. 2023 Aug;75(4):471-478. doi: 10.23736/S2724-6051.23.05270-9. Epub 2023 Jun 14. PMID 37314812
- [Background] Bertolo R, Iacovelli V, Cipriani C, Carilli M, Vittori M, Antonucci M, Maiorino F, Signoretti M, Petta F, Travaglia S, Panei M, Bove P. Ejaculatory function following transperineal laser ablation vs TURP for benign prostatic obstruction: a randomized trial. BJU Int. 2023 Jul;132(1):100-108. doi: 10.1111/bju.16008. Epub 2023 Mar 30. PMID 36917033
- [Background] Patelli G, Ranieri A, Paganelli A, Mauri G, Pacella CM. Transperineal Laser Ablation for Percutaneous Treatment of Benign Prostatic Hyperplasia: A Feasibility Study. Cardiovasc Intervent Radiol. 2017 Sep;40(9):1440-1446. doi: 10.1007/s00270-017-1662-9. Epub 2017 May 4. PMID 28474112
- [Background] Pacella CM, Patelli G, Iapicca G, Manenti G, Perretta T, Ryan CP, Esposito R, Mauri G. Transperineal laser ablation for percutaneous treatment of benign prostatic hyperplasia: a feasibility study. Results at 6 and 12 months from a retrospective multi-centric study. Prostate Cancer Prostatic Dis. 2020 Jun;23(2):356-363. doi: 10.1038/s41391-019-0196-4. Epub 2019 Dec 11. PMID 31827239
- [Background] Manenti G, Perretta T, Calcagni A, Ferrari D, Ryan CP, Fraioli F, Meucci R, Malizia A, Iacovelli V, Agro EF, Floris R. 3-T MRI and clinical validation of ultrasound-guided transperineal laser ablation of benign prostatic hyperplasia. Eur Radiol Exp. 2021 Sep 17;5(1):41. doi: 10.1186/s41747-021-00239-9. PMID 34532768
- [Background] Frego N, Saita A, Casale P, Diana P, Contieri R, Avolio PP, Lazzeri M, Hurle R, Buffi NM, Guazzoni GF, Lughezzani G. Feasibility, safety, and efficacy of ultrasound-guided transperineal laser ablation for the treatment of benign prostatic hyperplasia: a single institutional experience. World J Urol. 2021 Oct;39(10):3867-3873. doi: 10.1007/s00345-021-03685-7. Epub 2021 Apr 3. PMID 33811512
- [Background] de Rienzo G, Lorusso A, Minafra P, Zingarelli M, Papapicco G, Lucarelli G, Battaglia M, Ditonno P. Transperineal interstitial laser ablation of the prostate, a novel option for minimally invasive treatment of benign prostatic obstruction. Eur Urol. 2021 Jul;80(1):95-103. doi: 10.1016/j.eururo.2020.08.018. Epub 2020 Aug 28. PMID 32868137
- [Background] Cai HJ, Fang JH, Kong FL, Xu CK, Chen CH, Wang W, Huang B. Ultrasound-guided transperineal laser ablation for percutaneous treatment of benign prostatic hyperplasia: a new minimally invasive interventional therapy. Acta Radiol. 2022 Apr;63(4):553-558. doi: 10.1177/02841851211003289. Epub 2021 Mar 28. PMID 33779301